CLINICAL TRIAL: NCT00520026
Title: Suicide Prevention by Lithium - the Lithium Intervention Study
Acronym: SUPLI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: number of enrolled individuals after 5 years still off the estimated sample size
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Sanofi (Industry); Technische Universität Dresden (Other); University of Bonn (Other); Charite University, Berlin, Germany (Other); University of Erlangen-Nürnberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FKZ 01 GI9920 / 01 GI0220
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Suicide; Depressive Disorders
Keywords: suicide; prevention; lithium; suicidality
MeSH Terms: conditions — Suicide; Depressive Disorder; Suicidal Ideation | interventions — Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Lithium treatment
  Interventions: Drug: lithium
- 2 (Placebo Comparator): Placebo treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lithium
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The purpose of this study is to examine the proposed suicide preventive effects of lithium in a randomized controlled trial within a group of individuals with depressive disorders. The hypothesis being tested is that lithium treatment will significantly reduce the risk for another suicide attempt.

DETAILED DESCRIPTION:
Several studies have shown that there is a significantly increased risk of suicide related mortality in patients with a positive history of suicide attempts. This study is the first prospective, randomized, double-blind, placebo controlled multi-center trial focussing on the proposed suicide preventive effects of lithium in patients with suicidal behavior but not suffering from bipolar disorder or recurrent major depressive disorder. Patients with a recent history of a suicide attempt are treated with lithium or placebo during a 12 month-period. The hypothesis is that lithium treatment will lead to a 50 % reduction of suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

* suicide attempt within 3 months prior to the first drug administration
* occurrence of suicide attempt within the context of an affective spectrum disorder
* minimum age of 18 years
* ability to complete screening and baseline assessment
* ability to understand and provide informed consent

Exclusion Criteria:

* diagnosis of schizophrenia, borderline personality disorder, substance related disorders
* indication for long-term lithium treatment
* thyroid disease
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2001-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
occurrence of attempted and completed suicides | follow-up period of 1 year

SECONDARY OUTCOMES:
Specific aspects of the suicide attempt/completed suicide | follow-up period of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Hohagen, Prof., Study Director — Department of Psychiatry and Psychotherapy, Universitätsklinikum Schleswig-Holstein, Campus Luebeck; Bruno Müller-Oerlinghausen, Prof., Study Chair — Former Research Group Clinical Psychopharmacology, Department of Psychiatry and Psychotherapy, Charité-Universitätsmedizin Berlin, Campus Benjamin Franklin; Werner Felber, Prof., Study Chair — Department of Psychiatry and Psychotherapy, Medizinische Fakultät der Technischen Universität Dresden; Bernd Ahrens, PD, Study Chair — Department of Psychiatry and Psychotherapy, Universitätsklinikum Schleswig-Holstein, Campus Luebeck; Erik Lauterbach, Dr., Principal Investigator — Department of Psychiatry and Psychotherapy, Universitätsklinikum Schleswig-Holstein, Campus Luebeck; Thomas Bronisch, Prof., Study Chair — Max-Planck-Institute of Psychiatry Munich
Locations (5):
- Germany (5):
  - Department of Psychiatry and Psychotherapy, Charité-Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Department of Psychiatry and Psychotherapy, Rheinische Friedrich-Willhelms-Universität, Bonn
  - Department of Psychiatry and Psychotherapy, Medizinische Fakultät der Technischen Universität Dresden, Dresden
  - Department of Psychiatry and Psychotherapy, Universitätsklinikum Schleswig-Holstein, Campus Luebeck, Lübeck
  - Department of Psychiatry and Psychotherapy, Klinikum Nuremberg Nord, Nuremberg

REFERENCES:
- [Background] Lauterbach E, Ahrens B, Felber W, Oerlinghausen BM, Kilb B, Bischof G, Heuser I, Werner P, Hawellek B, Maier W, Lewitzka U, Pogarell O, Hegerl U, Bronisch T, Richter K, Niklewski G, Broocks A, Hohagen F. Suicide prevention by lithium SUPLI--challenges of a multi-center prospective study. Arch Suicide Res. 2005;9(1):27-34. doi: 10.1080/13811110590512886. PMID 16040577
- [Background] Muller-Oerlinghausen B, Felber W, Berghofer A, Lauterbach E, Ahrens B. The impact of lithium long-term medication on suicidal behavior and mortality of bipolar patients. Arch Suicide Res. 2005;9(3):307-19. doi: 10.1080/13811110590929550. PMID 16020173
- [Background] Muller-Oerlinghausen B, Berghofer A, Ahrens B. The antisuicidal and mortality-reducing effect of lithium prophylaxis: consequences for guidelines in clinical psychiatry. Can J Psychiatry. 2003 Aug;48(7):433-9. doi: 10.1177/070674370304800702. PMID 12971012
- [Background] Ahrens B, Muller-Oerlinghausen B. Does lithium exert an independent antisuicidal effect? Pharmacopsychiatry. 2001 Jul;34(4):132-6. doi: 10.1055/s-2001-15878. PMID 11518473